CLINICAL TRIAL: NCT00073554
Title: A Phase 2, Multicenter, Open-Label, Dose-Escalation Study to Evaluate the Safety and Activity of Alfimeprase in Patients With Acute Peripheral Arterial Occlusion
Brief Title: Alfimeprase for Thrombolysis in Acute Peripheral Arterial Occlusion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ARCA Biopharma, Inc. (Industry)
Collaborators: Premier Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HA002; NAPA-1
Record Dates: First submitted 2003-11-24; First posted 2003-11-26 (Estimated); Last update posted 2009-12-17 (Estimated); Status verified 2006-11

CONDITIONS: Arterial Occlusive Diseases; Peripheral Vascular Diseases; Thrombosis
MeSH Terms: conditions — Arterial Occlusive Diseases; Peripheral Vascular Diseases; Thrombosis | interventions — alfimeprase

INTERVENTIONS:
Drug: Alfimeprase

SUMMARY:
This trial is for patients with acute occlusion of one of the arteries supplying blood to the leg. The trial is designed to determine the safety and activity of a novel clot dissolving (thrombolytic) drug (alfimeprase).

ELIGIBILITY:
* Patients with acute peripheral arterial occlusion of the lower limb (onset of symptoms within 14 days)
* Rutherford Class I or IIa (minimal sensory loss, no muscle weakness, audible venous flow)
* Age 18 or above
* Able to consent
* Able to follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2003-06

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

REFERENCES:
- [Background] Toombs CF. Alfimeprase: pharmacology of a novel fibrinolytic metalloproteinase for thrombolysis. Haemostasis. 2001 May-Dec;31(3-6):141-7. doi: 10.1159/000048057. PMID 11910179